CLINICAL TRIAL: NCT04079036
Title: Decision Support System for Anesthetists for In-room Monitoring of the Level of Consciousness, Neuro-muscular Blocking and Nociception Employing Data Fusion and Artificial Intelligence
Brief Title: Decision Support System for Anesthetists
Acronym: Serenity
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: University of Sao Paulo (Other); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Joaquim Edson Vieira, Phd Anesthesiology Professor and Principal invesigator, University of Sao Paulo General Hospital
Other Study IDs: CAAE 03424918.6.0000.0068
Record Dates: First submitted 2019-07-10; First posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Anesthesia
Keywords: General Anesthesia; Anesthesia Awareness; Anesthesia overdose
MeSH Terms: conditions — Intraoperative Awareness

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (12):
- Underweight Adult Male: Male patients with Underweight BMI classification and more than 20 years old https://www.cdc.gov/healthyweight/assessing/bmi/adult_bmi/index.html
- Healthy Weight Adult Male: Male patients with Healthy Weight BMI classification and more than 20 years old
- Overweight Adult Male: Male patients with OverWeight or Obese BMI classification and more than 20 years old
- Underweight Adult Female: Female patients with Underweight BMI classification and more than 20 years old
- Healthy Weight Adult Female: Female patients with Healthy Weight BMI classification and more than 20 years old
- Overweight Adult Female: Female patients with Overweight or Obese BMI classification and more than 20 years old
- Underweight children Male: Male patients less than 20 year old, and with Underweight BMI classification https://www.cdc.gov/healthyweight/assessing/bmi/childrens_bmi/about_childrens_bmi.html
- Healthy Weight children Male: Male patients less than 20 year old, and with Healthy Weight BMI classification
- Overweight children Male: Male patients less than 20 year old, and with Overweight or Obese BMI classification
- Underweight children Female: Male patients less than 20 year old, and with Underweight BMI classification https://www.cdc.gov/healthyweight/assessing/bmi/childrens_bmi/about_childrens_bmi.html
- Healthy Weight children Female: Female patients less than 20 year old, and with Overweight or Obese BMI classification
- Overweight children Female: Female patients less than 20 year old, and with Overweight or Obese BMI classification

SUMMARY:
The balanced anesthesia process contains three main parts: the control of hypnosis, analgesia, and neuromuscular blockade. For the induction phase, the anesthesiologist performs protocols based on prior planning specific to each patient and usually performs these controls by monitoring the classic vital signs and other clinical signs for the maintenance phase.

In a way, this professional is the controller in a control system that acts on the plant (the patient) through the infusion of hypnotic drugs, analgesics and neuromuscular blockers. In addition, the anesthesiologist estimates the state of consciousness, the level of analgesia and the level of neuromuscular blockage through other indirect measures, as well as a state observer.

There are different techniques for direct monitoring of these three anesthesia variables (DoA, NMB and NoL), such as BIS and Narcotrend, but all have some disadvantages, especially when the anesthesia process combines different drugs. This work proposes a new way of evaluating DoA, NMB and NoL using data fusion techniques to combine classical clinical signs with advanced EEG monitoring techniques to provide a decision support system for the anesthesiologist.

DETAILED DESCRIPTION:
The balanced anesthesia process contains three main parts: the control of hypnosis, the analgesia and neuromuscular blockade. For the induction phase, the anesthesiologist performs protocols based on prior planning specific to each patient. Normally, the anesthesiologist controls the process by monitoring the classical vital signs and other clinical most common signs during the maintenance phase. In a way, this professional is the controller in a control system that acts on the plant (the patient) through the infusion of hypnotic and analgesic drugs and neuromuscular blockers.

In addition, the anesthesiologist estimates the the level of consciousness, of nociception and the level of neuromuscular blockade through these indirect measurements, just as a state observer in a control system would do.

There are different techniques for the direct monitoring of these three variables of anesthesia (DoA, NMB and NoL), such as BIS and Narcotrend, but all of them present a few disadvantages and mis-measurements, especially when the anesthesia process combines different drugs.

This work proposes a new way of evaluating DoA, NMB and NoL, using techniques to combine classical clinical signs with advanced EEG monitoring, to provide a decision support system for the anesthesiologist.

For this, we will perform data acquisition from the equipment usually used in surgical procedures with general anesthesia, such as ECG, EEG, blood pressure, mechanical ventilation, among others.

In short, all data of the patient's vital signs during the procedure and the actions taken by the anesthesiologist and surgeons.

The data will be concentrated on a specific equipment, and will be analyzed together with the data of other patients to improve the mathematical models involved in the process.

ELIGIBILITY:
Inclusion Criteria:

* Patients under general anesthesia

Exclusion Criteria:

* Cerebral Palsy patients

Ages: 1 Month to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing surgical procedures with general anesthesia
Sampling Method: Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Heart Rate | 2 to 3 months of different surgical procedures
  HR - Heart Rate - unit: [bpm], will be stored in real time during the surgical procedure.
Arterial blood pressure | 2 to 3 months of different surgical procedures
  P_INV - Invasive blood pressure - unit: [mmHg], will be stored in real time during the surgical procedure.
Mean Arterial Pressure | 2 to 3 months of different surgical procedures
  MAP - Mean Arterial Pressure - unit: [mmHg], will be stored in real time during the surgical procedure.
Non Invasive Blood pressure | 2 to 3 months of different surgical procedures
  P_NINV - Non Invasive blood pressure - unit: [mmHg/mmHg], will be stored in real time during the surgical procedure.
Conscience Level | 2 to 3 months of diferent surgical procedures
  CL - Consciousnesses Level (through BIS) - unit: [u 0-100] will be stored in real time during the surgical procedure.
Inspired anesthetic concentration | 2 to 3 months of different surgical procedures
  FiAA - Inspired fraction of anesthetic agent - unit: [% of Volume], will be stored in real time during the surgical procedure.
Inspired carbon dioxide concentration | 2 to 3 months of different surgical procedures
  FiCO2 - CO2 inspired Fraction - unit: [% of Volume], will be stored in real time during the surgical procedure.
Inspired Nitrous Oxide concentration | 2 to 3 months of different surgical procedures
  FiN2O - N2O inspired Fraction - unit: [% of Volume], will be stored in real time during the surgical procedure.
Blood oxygen saturation | 2 to 3 months of different surgical procedures
  SpO2 - Peripheral capillary oxygen saturation - unit: [%], will be stored in real time during the surgical procedure.
Exhaled Carbon Dioxide concentration | 2 to 3 months of different surgical procedures
  EtCO2 - End-tidal CO2 concentration (CO2 Exhaled Fraction) - unit: [% of Volume], will be stored in real time during the surgical procedure.
Exhaled Anesthetic concentration | 2 to 3 months of different surgical procedures
  EtAA - Anesthetic agents Exhaled Fraction - unit: [% of Volume], will be stored in real time during the surgical procedure.
Anesthetic agent infusion rate | 2 to 3 months of different surgical procedures
  IR_Anes - Infusion Rate of anesthetic agent - unit: [mg/hr], will be stored in real time during the surgical procedure.
Analgesic agent infusion rate | 2 to 3 months of different surgical procedures
  IR_Analg - Infusion rate of Analgesic agent - unit: [mg/hr], will be stored in real time during the surgical procedure.
Neuro-muscular Block agent infusion rate | 2 to 3 months of different surgical procedures
  IR_NMB - Infusion rate of neuro-muscular block agent - unit: [mg/hr], will be stored in real time during the surgical procedure.
Ventilation respiratory rate | 2 to 3 months of different surgical procedures
  RR - Respiratory Rate - unit: [bpm], will be stored in real time during the surgical procedure.
Ventilation Tidal volume | 2 to 3 months of different surgical procedures
  Vt - Tidal Volume - unit: [mL], will be stored in real time during the surgical procedure.
Ventilation Minute Volume | 2 to 3 months of different surgical procedures
  Vm - Minute Volume - unit: [L/min], will be stored in real time during the surgical procedure.
Ventilation maximum pressure per cycle | 2 to 3 months of different surgical procedures
  Pmax - Maximum pressure during the inspiration cycle - unit: [cmH2O], will be stored in real time during the surgical procedure.
Ventilation Plateau pressure | 2 to 3 months of different surgical procedures
  Pplateau - Plateau pressure during the inspiration cycle - unit: [cmH2O], will be stored in real time during the surgical procedure.
Ventilation PEEP | 2 to 3 months of different surgical procedures
  PEEP - Positive end of expiration pressure - unit: [cmH2O], will be stored in real time during the surgical procedure.
Primary anesthesia Data - related to the manual infusion of drugs | 2 to 3 months of different surgical procedures
  Every monitored clinical variable, related to the manual infusion of drugs, will be stored in real time during the surgical procedure.
  Every infusion made manually by the anesthesiologist during the procedure should be recorded, always considering the total amount infused and the time it occurred.
Preoperative patient medical records - General state of the patient in ASA. | 2 to 3 months of different surgical procedures
  Anesthesia related preoperative information from the patient, such as prior use of opioids, ASA and METS indexes.
  ASA - Physical state of the patient - unit: [u] P1 to P5
Preoperative patient medical records - General state of the patient in METS. | 2 to 3 months of different surgical procedures
  Anesthesia related preoperative information from the patient, such as prior use of opioids, ASA and METS indexes.
  METS - Functional state of the patient - unit: [u]
Preoperative patient medical records - Clinical state of the patient - Age | 2 to 3 months of different surgical procedures
  Anesthesia related preoperative information from the patient, such as:
  I - Age - unit: [years]
Preoperative patient medical records - Clinical state of the patient - gender | 2 to 3 months of different surgical procedures
  Anesthesia related preoperative information from the patient, such as:
  G - Gender - unit: Male or Female
Preoperative patient medical records - Clinical state of the patient - Weight | 2 to 3 months of different surgical procedures
  Anesthesia related preoperative information from the patient, such as:
  P - Weight - unit: [Kg]
Preoperative patient medical records - Clinical state of the patient - Height | 2 to 3 months of different surgical procedures
  Anesthesia related preoperative information from the patient, such as:
  A - Height - unit: [cm]

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim E Vieira, MD, PhD, Principal Investigator — University of Sao Paulo School of Medicine
Locations (1):
- Hospital das Clínicas - Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schnider TW, Minto CF, Struys MM, Absalom AR. The Safety of Target-Controlled Infusions. Anesth Analg. 2016 Jan;122(1):79-85. doi: 10.1213/ANE.0000000000001005. PMID 26516801
- [Background] Karl J Åström, Björn Wittenmark. Computer-Controlled Systems: Theory and Design. Dover Books on Electrical Engineering. ISBN: 0486284042. Courier Corporation, 2013
- [Result] Ahmad AM. Recent advances in pharmacokinetic modeling. Biopharm Drug Dispos. 2007 Apr;28(3):135-43. doi: 10.1002/bdd.540. PMID 17295411
- [Result] Iselin-Chaves IA, Flaishon R, Sebel PS, Howell S, Gan TJ, Sigl J, Ginsberg B, Glass PS. The effect of the interaction of propofol and alfentanil on recall, loss of consciousness, and the Bispectral Index. Anesth Analg. 1998 Oct;87(4):949-55. doi: 10.1097/00000539-199810000-00038. PMID 9768800